CLINICAL TRIAL: NCT02595957
Title: Genomic Services Research Program
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160017; 16-HG-0017
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-02

CONDITIONS: Colon Cancer; Breast Cancer
Keywords: Genome Sequencing; Secondary Findings; Return of Results; Natural History; Exome Sequencing
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cascade Testing: Family members of individuals who have received secondary genomic findings after exome/genome sequencing
- Secondary findings recipients: Individuals who have received secondary genomic findings after exome/genome sequencing

SUMMARY:
Background:

Genes are the instructions a person s body uses to function. Genome sequencing reads through all of a person s genes. Everyone has many gene variants, and most do not cause disease. Some gene variants called secondary findings may be important for a person s health even if they are not related to the reason why a person had genome sequencing done. Researchers want to learn more about what it means to have a secondary finding.

Objectives:

To learn about how gene variants may affect a person s health.

To learn about how people understand their genetic test results.

Eligibility:

People with secondary findings from genetic testing done as part of a research study, clinical care, or other methods.

Design:

Participants may be asked to do an online survey and phone interview to ask what they think about their results, their healthcare, and if they talk with their family about the result.

Eligible participants may be offered a visit to the NIH Clinical Center where they will be evaluated for health problems related to the secondary finding.

DNA samples that were already collected may be studied.

Participants may be asked to send in a second DNA sample (blood or saliva). These will be used to verify any findings.

Participants who have a secondary finding can get genetic counseling.

DETAILED DESCRIPTION:
The implementation of genome and exome sequencing creates challenges and opportunities, particularly with respect to the return of medically-actionable secondary findings (SF). This study seeks to investigate the utility and effectiveness of returning SF generated via research or clinical sequencing by studying individuals who have received such findings. Our objectives with this protocol have evolved over time and have been substantially informed by our experiences in returning SF through sequencing initiatives such as the ClinSeq(R) study, the Clinical Center Genomics Opportunity (CCGO), and the Secondary Genomic Findings Service (SGFS). Our work with these studies/initiatives suggests that much remains unknown about how recipients of SF understand these findings, communicate them to their health professionals and families, and whether they adhere to recommended health-preserving actions in both the short and long-term. As well, recipients of SF are an unselected population in which to investigate penetrance of disorders associated with SF genes. Thus, this protocol aims to explore important questions of clinical utility associated with SF return and penetrance of SF-related disorders. Healthcare actions and family communication (clinical utility) are assessed by interviews and surveys with SF recipients. This protocol also includes a pilot program in which selected participants will be invited to the NIH for bespoke phenotyping to uncover the presence of disease and explore avenues to develop interventions to enhance outcomes.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

We employ a referral form through SurveyMonkey to receive referrals from recruitment partners or self-referrals. This serves as an intake form and self-reported eligibility review. This form asks for contact information, key information about the prospective participant s SF,

and subjective understanding of their result.

If we conclude, based on a review of the SF and available personal and/or family history, that the pathogenicity of the SF is not at least likely pathogenic, that participant may be eligible for the survey, interview, and/or re-contact for future follow-up, but will not complete any other protocol procedures (such as cascade testing). If a participant is consented and information arises during the social and behavioral study procedures that lead study staff to believe the genetic result does not qualify as an SF, the participant will be

considered a screen failure and will not continue with study procedures.

We plan to offer enrollment in this protocol to English- or Spanish-speaking recipients of SF. We do not have trained staff who can conduct the interviews in languages other than English and Spanish.

If a caregiver of a minor or adult who is unable to consent is enrolled as an index participant to complete the survey and interview on behalf of the SF recipient, they may also be eligible for cascade testing to relate presence of an SF-related phenotype in a family member with presence or absence of SF genotype.

-We may enroll a child in this protocol if he/she is the only person in his/her family who has the SF, is symptomatic of the disease, or is in the age range to receive screening for the disease (e.g., Wilson disease and familial hypercholesterolemia have childhood onset).

We will not enroll neonates (less than one month old).

* We may enroll adults who are unable to consent (i.e., an individual who is impaired at the time of consent) in this protocol if he/she is the only person in his/her family who has the SF, is symptomatic of the disease, or is in the age range to receive screening for the disease.
* We may enroll women who are pregnant in this protocol and women who become pregnant during the study can continue their participation. We will not perform prenatal genetic testing.
* NIH staff members are not prohibited from enrollment if they meet the study s eligibility criteria. The study team will make every effort to protect the confidentiality of the NIH staff member s health information, to minimize any pressure on or discomfort of the NIH staff

member and provide a copy of the NIH Frequently Asked Questions (FAQs) for Staff Who are Considering Participation in NIH Research , before consent is obtained.

Ages: 1 Month to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have participated in a sequencing study at the NIH or elsewhere who have have received secondary findings through other means are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-09-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Health impacts of SF receipt | enrollment and return of results
  We will assess the health impacts of SF receipt and healthcare processes affecting outcomes in SF recipients.
Adherence to medical recommendations | enrollment and return of results
  We will assess what individual, community, and systemic factors influence recipients' follow through on recommendations and how they communicate SF results with family members.
Family based positive predictive value | return of results and cascade testing
  We will assess penetrance using the family-based positive predictive value metric
Responses and perceptions | enrollment and return of results
  We will assess affective responses and healthcare and behavioral changes to receiving positive SF results

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sapp JC, Johnston JJ, Driscoll K, Heidlebaugh AR, Miren Sagardia A, Dogbe DN, Umstead KL, Turbitt E, Alevizos I, Baron J, Bonnemann C, Brooks B, Donkervoort S, Jee YH, Linehan WM, McMahon FJ, Moss J, Mullikin JC, Nielsen D, Pelayo E, Remaley AT, Siegel R, Su H, Zarate C; NISC Comparative Sequencing Program; Manolio TA, Biesecker BB, Biesecker LG. Evaluation of Recipients of Positive and Negative Secondary Findings Evaluations in a Hybrid CLIA-Research Sequencing Pilot. Am J Hum Genet. 2018 Sep 6;103(3):358-366. doi: 10.1016/j.ajhg.2018.07.018. Epub 2018 Aug 16. PMID 30122538
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-HG-0017.html